CLINICAL TRIAL: NCT06094439
Title: Targeted Metabolomics of Spent Embryo Culture Medium
Brief Title: Targeted Metabolomics and Spent Embryo Culture Medium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: gyn-medicum Göttingen (Other)
Responsible Party: Sponsor
Other Study IDs: gyn-medicumGöttingen
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Embryo Culture Media; Metabolomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 50 µl of spent embryo culture media
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good or poor embryo quality: morphological evaluation will be performed by an expert embryologist to confirm poor and good embryo quality
- metabolomics profiles: metabolomics profiles will be performed by a Metabolomics core facility

SUMMARY:
More than 8 million babies have been born through in vitro fertilization (IVF). Non-invasive observation of embryos in vitro to better understand their development is becoming increasingly important. Morphology has been used as standard from the beginning, but has the disadvantage of subjectivity. Now the emphasis in basic and clinical research is on developing rapid, quantitative, non-invasive tests. Hence comes the idea of metabolic profiling of spent embryo culture medium (SECM) as a biomarker. This could be useful for understanding and improving the nutritional environment of oocytes and embryos. The goal of our study is to determine metabolic profiles of the SECM in combination with morphological assessments to better understand the nutritional requirements of the embryo. The goal would be to optimize media specifically, depending on patient and embryo characteristics ("personalized medicine") ("the embryo in vitro as patient").

DETAILED DESCRIPTION:
Following successful fertilization (day 1), each embryo will be cultured for 5-6 days (day 5-6) to form the blastocyst. Then, morphological evaluation will be performed by an expert embryologist to confirm poor and good embryo quality. At the end of the culture, 50 µl of SECM will be collected from each embryo and stored for metabolomics analysis. Samples including medium only and no embryos will be used as controls. The metabolome will be characterized in SECM samples using the respective assay targeted kit.

ELIGIBILITY:
Inclusion Criteria:

- Available spent embryo culture medium (SECM) samples with Informed consent

Exclusion Criteria:

* Diabetes

Ages: 35 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The available spent embryo culture medium (SECM) samples (n> 50 samples) will be collected from embryos produced by IVF and ICSI during nine months. The experimental groups will include: I) SECM obtained from good quality embryos and II) SECM obtained from poor quality embryos. In this study, the samples are classified according to their morphological characteristics of embryos, BMI and age of the women.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Metabolomics profiles of good vs. Metabolomics profiles of poor quality embryos | 24 months
  The metabolome will be characterized in SECM samples of good and poor quality embryos using the respective assay kit. This method needs to be developed and analyses are planned in cooperation with the metabolomics core facility; the targeted metabolomics approach using the MxP® Quant 500 kit assay (BIOCRATES Life Sciences AG, Innsbruck, Austria) will be used. The kit plates are used for the quantification of amino acids, acylcarnitines, sphingomyelins, phosphatidylcholines, hexoses, and biogenic amines in SECM of good and poor quality embryos. Results of metabolic set enrichment analysis (MSEA) and metabolic pathway analysis (MetPA) will be used as the final results to compare the metabolite profiles of good and poor quality embryos .

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schmutzler, PD Dr. med., Study Chair — gyn-medicum Göttingen
Locations (1):
- Gyn-Medicum, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Current study dose not contain any individual person's data in any form (including any individual details, images or videos).

REFERENCES:
- [Background] Inoue N, Nishida Y, Harada E, Sakai K, Narahara H. GC-MS/MS analysis of metabolites derived from a single human blastocyst. Metabolomics. 2021 Jan 25;17(2):17. doi: 10.1007/s11306-021-01770-x. PMID 33495963
- [Background] Siristatidis C, Dafopoulos K, Papapanou M, Stavros S, Pouliakis A, Eleftheriades A, Sidiropoulou T, Vlahos N. Why Has Metabolomics So Far Not Managed to Efficiently Contribute to the Improvement of Assisted Reproduction Outcomes? The Answer through a Review of the Best Available Current Evidence. Diagnostics (Basel). 2021 Sep 2;11(9):1602. doi: 10.3390/diagnostics11091602. PMID 34573944
- [Background] Cimadomo D, Rienzi L, Conforti A, Forman E, Canosa S, Innocenti F, Poli M, Hynes J, Gemmell L, Vaiarelli A, Alviggi C, Ubaldi FM, Capalbo A. Opening the black box: why do euploid blastocysts fail to implant? A systematic review and meta-analysis. Hum Reprod Update. 2023 Sep 5;29(5):570-633. doi: 10.1093/humupd/dmad010. PMID 37192834